CLINICAL TRIAL: NCT01059201
Title: Exome Sequencing in Autistic Spectrum Disorder Patients With Altered Cholesterol Homeostasis
Brief Title: Exome Sequencing in Autistic Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100022; 10-CH-0022
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-05-15

CONDITIONS: Autism Spectrum Disorder; Autism; Autistic Disorder
Keywords: Autism Spectrum Disorder; Cholesterol; Exome Sequencing; Autistic Spectrum Disorder; ASD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
Background:

* Research into the genetic causes of autism spectrum disorder (ASD) involves studies of the DNA of children with autism. New DNA sequencing technology allows researchers to study specific genes in search of genetic changes that may cause or contribute to ASD. Individuals who donated DNA to the Autism Genetic Resource Exchange may benefit from further study of their DNA samples with more advanced DNA sequencing technology.
* The role of cholesterol in individuals with ASD is currently under investigation. Research has suggested that abnormal cholesterol levels in children with autism may be related to genetic mutations or changes in how cholesterol is regulated in the body.

Objectives:

- To study existing blood samples of children with autism spectrum disorders to evaluate the relationship between genetic traits and cholesterol function.

Eligibility:

- Children with ASD who donated blood samples to the Autism Genetic Resource Exchange.

Design:

* Parents/guardians of minor children with ASD will provide consent for further research to be performed on existing DNA samples in the Autism Genetic Research Exchange databank. Information from this research may be provided to the consenting parents/guardians on a case by case basis, as directed by the researchers.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder characterized by functional deficits in three domains: social interaction, communication, and stereotypic behavior. Prevalence has been estimated to be approximately 1/166 children and the public health impact is significant. ASD clearly has a genetic component; however, identification of specific etiologies has been complicated by the heterogeneous nature of ASD. One approach to minimize this problem is to define endophenotypes that can subcategorize ASD patients. Based on our work with Smith-Lemli-Opitz syndrome, we have investigated whether alterations in cholesterol homeostasis may contribute to ASD. We found in 200 ASD subjects that 23% of subjects had serum cholesterol levels less than or equal to 2.28th centile and 9% had levels greater than or equal to 97.72nd centile. Analysis of the sterol profile suggested that the hypocholesterolemia was due to a synthetic defect rather than decreased oral intake. Thus we hypothesize that ASD patients with abnormal cholesterol levels will have polymorphisms or mutations of either genes involved in cholesterol homeostasis or genes encoding proteins whose function is altered by changes in cholesterol levels. To test this hypothesis we propose to 1) use serum cholesterol levels to define ASD endophenotypes and 2) to perform genomic resequencing of all known exons in hypo- and normocholesterolemic ASD patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Prior participation in Autism Genetic Research Exchange
  2. Multiple affected children with ASD
  3. Willingness to contact the NIH and reconsent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2010-01-21; Study Completion 2017-05-15

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (3):
- United States (3):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Newschaffer CJ, Croen LA, Daniels J, Giarelli E, Grether JK, Levy SE, Mandell DS, Miller LA, Pinto-Martin J, Reaven J, Reynolds AM, Rice CE, Schendel D, Windham GC. The epidemiology of autism spectrum disorders. Annu Rev Public Health. 2007;28:235-58. doi: 10.1146/annurev.publhealth.28.021406.144007. PMID 17367287
- [Background] Jacobson JW, Mulick JA. System and cost research issues in treatments for people with autistic disorders. J Autism Dev Disord. 2000 Dec;30(6):585-93. doi: 10.1023/a:1005691411255. PMID 11261469
- [Background] Seltzer MM, Shattuck P, Abbeduto L, Greenberg JS. Trajectory of development in adolescents and adults with autism. Ment Retard Dev Disabil Res Rev. 2004;10(4):234-47. doi: 10.1002/mrdd.20038. PMID 15666341